CLINICAL TRIAL: NCT07018141
Title: Clinical And Digital Evaluation Of Wear Resistance Of Bioactive Pits And Fissure Sealant With And Without Etching Versus Conventional Resin Based Pits And Fissure Sealants: A RANDOMIZED CLINICAL TRIAL
Brief Title: Wear Resistance Of Bioactive With And Without Etching Vs. Conventional Resin-Based Fissure Sealants
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Cairo University (Other)
Responsible Party: Principal Investigator, Rana hossam eldin mahfouz, Master degree student dentist, Cairo University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: Operative 4
Record Dates: First submitted 2025-05-21; First posted 2025-06-12 (Actual); Last update posted 2025-06-12 (Actual); Status verified 2025-06

CONDITIONS: Pit and Fissure Caries
Keywords: Pit and Fissure Caries
MeSH Terms: conditions — Van der Woude syndrome | interventions — Pit and Fissure Sealants

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Fluoride Releasing bioactive Pit and Fissure Sealant with etchant (Experimental): Fluoride Releasing bioactive Pit and Fissure Sealant with etchant application.
  Interventions: Other: Bioactive Sealant with Etching: Participants in this group received a fluoride-releasing bioactive pit and fissure sealant (BeautiSealant, Shofu) applied after etching the tooth surface with 37% phosp
- Fluoride Releasing bioactive Pit and Fissure Sealant without etchant (Experimental): Fluoride Releasing bioactive Pit and Fissure Sealant without etchant application.
  Interventions: Other: Bioactive Sealant without Etching: In this group, the same bioactive sealant (BeautiSealant, Shofu) was applied directly without acid etching. This simplified technique evaluates the sealant's effecti
- conventional resin based pits and fissure sealant (Active Comparator): Conventional resin-based sealant with etchant application
  Interventions: Other: Conventional Resin-Based Sealant with Etching (Control): This group received a conventional resin-based sealant (Fisseal, Promedica) following standard acid etching. This technique represents the trad

INTERVENTIONS:
Other: Bioactive Sealant with Etching: Participants in this group received a fluoride-releasing bioactive pit and fissure sealant (BeautiSealant, Shofu) applied after etching the tooth surface with 37% phosp — This group received BeautiSealant (a bioactive giomer-based sealant) applied after etching the enamel surface with 37% phosphoric acid for 15 seconds. The etching process creates micro-retentive patterns in the enamel to enhance micromechanical bonding, potentially improving the sealant's retention and wear resistance while also benefiting from the bioactive material's fluoride release and enamel remineralization properties.
  Arms: Fluoride Releasing bioactive Pit and Fissure Sealant with etchant
Other: Bioactive Sealant without Etching: In this group, the same bioactive sealant (BeautiSealant, Shofu) was applied directly without acid etching. This simplified technique evaluates the sealant's effecti — In this group, BeautiSealant was applied directly to the tooth surface without prior etching. The goal was to simplify the procedure by eliminating the etching step, relying instead on the sealant's chemical bonding and bioactive properties (such as fluoride release and S-PRG technology) to maintain retention and resist wear, while reducing the risk of enamel alteration and improving clinical efficiency.
  Arms: Fluoride Releasing bioactive Pit and Fissure Sealant without etchant
Other: Conventional Resin-Based Sealant with Etching (Control): This group received a conventional resin-based sealant (Fisseal, Promedica) following standard acid etching. This technique represents the trad — This group served as the control and received Fisseal (a conventional resin-based sealant) applied following standard etching with 37% phosphoric acid. This method is considered the gold standard for fissure sealing, offering strong micromechanical adhesion and proven wear resistance, making it a reliable benchmark for evaluating the performance of newer bioactive materials.
  Arms: conventional resin based pits and fissure sealant

SUMMARY:
This randomized clinical trial aimed to compare the wear resistance and clinical performance of bioactive versus conventional resin-based pit and fissure sealants over a 12-month period. Conducted on young adults with sound, caries-susceptible molars, the study evaluated three groups: bioactive sealants applied with and without etching, and conventional resin-based sealants with etching. Clinical assessments and 3D digital scans were used to measure sealant retention and wear. The study seeks to determine whether bioactive sealants, especially when applied without etching, provide comparable long-term protection and durability to conventional sealants, potentially simplifying application without compromising effectiveness.

DETAILED DESCRIPTION:
This study is a randomized controlled clinical trial designed to evaluate and compare the wear resistance and clinical performance of bioactive pit and fissure sealants-applied with and without acid etching-against conventional resin-based sealants in young adults aged 18-25 with caries-susceptible, sound first permanent molars. Seventy-five teeth were randomly assigned to three groups: Group 1 received a bioactive giomer-based sealant (BeautiSealant) with etching, Group 2 received the same sealant without etching, and Group 3 received a conventional resin-based sealant (Fisseal Promedica) with etching. Sealant retention and wear were evaluated clinically using modified USPHS criteria and digitally using intraoral 3D scanning at baseline, 6 months, and 12 months. The aim was to determine if omitting the etching step in bioactive sealants compromises their effectiveness, offering a simpler yet reliable alternative to conventional methods. The findings are expected to guide clinical decision-making on the most efficient and durable sealant protocols for caries prevention.

ELIGIBILITY:
Inclusion Criteria:

* patients aged between 18-25 years old with caries susceptible sound fissures and good oral hygiene
* They should not show any signs of caries by visual tactile examination method and VistaProof fluoroscent camera
* Teeth should have intact contact with opposing teeth, no previous restorations in other surfaces, no previous sealing procedures and scoring 0.9 or less when tested and VistaProof.
* Medically free patients.

Exclusion Criteria:

* Patients with poor oral hygiene, lack of compliance, parafunctional habits, tempro-mandibular joint disorders, periodontal disease, severe medical conditions, allergic history concerning methacrylates, rampant caries, heavy smoking and xerostomia.
* Teeth with caries pits and fissures, developmental anomalies, periapical pathology or signs of pulpal pathology, hypersensitivity, possible prosthodontic restoration, heavy occlusion and occlusal contacts, history of bruxism, severe periodontal affection and scoring >0.9 when tested with VistaProof

Ages: 18 Years to 25 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 23 (Estimated)
Dates: Start 2025-08 (Estimated); Primary Completion 2025-09 (Estimated); Study Completion 2026-10 (Estimated)

PRIMARY OUTCOMES:
retention of wear resistance of the sealants | 3,6,9 and 12 months
  modified USPHS criteria

SECONDARY OUTCOMES:
quantitative wear assesment | 12 months
  digital scanner